CLINICAL TRIAL: NCT03041337
Title: Morphological and Functional Response of the Right Heart and Pulmonary Circulation
Brief Title: Right Heart International NETwork During Exercise in Different Clinical Conditions
Acronym: RIGHT-Net
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Responsible Party: Principal Investigator, Eduardo Bossone, Director of Cardiology and Coronary Care Unit, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Other Study IDs: RIGHT-Net
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Echocardiography, Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Cohort of patients referred to our echocardiography laboratory to work assessment procedures and without any cardiovascular risk factor. They will underwent stress echocardiography.
  Interventions: Diagnostic Test: stress echocardiography
- cardio-respiratory diseases: patients with any possible cardiovascular and respiratory condition. They will underwent stress echocardiography.
  Interventions: Diagnostic Test: stress echocardiography

INTERVENTIONS:
Diagnostic Test: stress echocardiography — stress echocardiography will be performed in accordance with the current guidelines on a variable load 45° cycle ergometer with an incremental workload of 25 W every 2 minutes up to the symptom-limited maximal tolerated workload. Echocardiographic measurements will be acquired at baseline, at peak exercise and during recovery of 5 minutes.
  The electrocardiogram and blood pressure will be monitored at each workload. Termination criteria and / or positive test criteria for inducible myocardial ischemia will follow the current recommendations

SUMMARY:
The aim of this registry will be to compare the pathophysiological response of the morphology and function of the right heart and pulmonary circulation assessed with resting and stress-echocardiography in patients with various cardiovascular diseases, to compare them to healthy individuals. The physiological response in healthy individuals as well as elite athletes, defined as athletes participating at national and international competitions, will also be evaluated. Patients will be enrolled both prospectively as well as retrospectively and the will be evaluated by resting and stress echocardiography, which are part of the routine clinical practice.

All clinical outcome measures will be collected as part of routine examinations. The measurements will include systolic and diastolic pump function of the right and left ventricles and other echocardiographic parameters. Moreover, a comparison of these parameters among different groups will be performed. Other optional assessments will include: exercise capacity assessed with 6-minute walking distance, World Health Organization functional class (WHO functional class), peak oxygen uptake assessed by spiroergometry. Patients will be evaluated at baseline and each year with the aforementioned procedures according to the sites clinical routine.

DETAILED DESCRIPTION:
Patients will be evaluated with a routinely performed resting and stress echocardiography. Moreover, physical examination and ECG will be performed and past medical history will be collected. Optional procedures comprise of quality of life assessment (SF-36 questionnaire), six minute walking distance (6MWD), cardiopulmonary exercise testing (CPET), routine laboratory including biochemical work-up.

Comparison among different cohorts of patients with regards to right heart morphology and function at rest, assessed during a routinely performed resting and stress echography. The following parameters will be evaluated:

* Right ventricular (RV) diameters
* RV free wall thickness
* End-diastolic and end-systolic left ventricular volumes and ejection fraction
* Right atrial (RA) area
* End-diastolic and end-systolic RV area and % shortening of the areas of the right ventricle
* Tricuspid regurgitation velocity (TRV) and severity
* Tricuspid annular plane systolic excursion (TAPSE)
* Inferior vena cava diameter and % of collapsibility
* TAPSE at peak exercise and after 5 minutes recovery
* TRV at peak exercise and after 5 minutes recovery
* RV end-diastolic and end-systolic area and % shortening of the areas at peak exercise and after 5 minutes recovery
* RA area at peak exercise and after 5 minutes recovery
* Left ventricular end-diastolic and end-systolic volume and ejection fraction at peak exercise and after 5 minutes recovery
* Left ventricular eccentricity index at peak exercise and after 5 minutes recovery

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males and females ≥ 18 years' old
* Ability to understand study-specific design and procedures and provide informed consent to the study

Exclusion Criteria:

* Inability to perform exercise stress test
* Active smoker
* Pregnancy and/or lactation
* Active malignancy
* End-stage renal disease requiring dialysis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy subjects will be enrolled both retrospectively as well as prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Right Ventricle contractile reserve | ten years
  Difference of tricuspid regurgitation velocity at rest to peak exercise (m/s)

SECONDARY OUTCOMES:
All-cause Mortality | ten years
  All cause of mortality
Cardiovascular Mortality | ten years
  all cardiovascular mortality
RV internal end-diastolic diameters | ten years
  measurement of basal and midcavity RV internal end-diastolic diameters from the four-chamber view in mm
tricuspid annular plane systolic excursion (TAPSE) | ten years
  tricuspid annular plane systolic excursion (TAPSE) determined in M-mode in mm

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bossone, Study Chair — Azienda Universitaria Ospedaliera "S. Giovanni e Ruggi d'Aragona"
Locations (1):
- Cardiology and Coronary Care Unit, Cava de' Tirreni, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Luca M, Ferrara F, Gargani L, Argiento P, Bandera F, Carbone A, Castaldo R, D'Agostino A, D'Alto M, D'Andrea A, D'Assante R, Franzese M, Giardino F, Grunig E, Kasprzak JD, Limongelli G, Passaro E, Pugliese NR, Rega S, Schiavo A, Vriz O, Wierzbowska-Drabik K, Cittadini A, Naeije R, Bossone E, Marra AM; RIGHT Heart International NETwork. Exercise Doppler Echocardiography of the Right Heart and Pulmonary Circulation in Patients With Cardiovascular Risk Factors: Observations From the RIGHT Heart International NETwork (RIGHT-NET). Chest. 2025 Dec;168(6):1460-1470. doi: 10.1016/j.chest.2025.06.020. Epub 2025 Jun 19. PMID 40543748
- [Derived] Gargani L, Pugliese NR, De Biase N, Mazzola M, Agoston G, Arcopinto M, Argiento P, Armstrong WF, Bandera F, Cademartiri F, Carbone A, Castaldo R, Citro R, Cocchia R, Codullo V, D'Alto M, D'Andrea A, Douschan P, Fabiani I, Ferrara F, Franzese M, Frumento P, Ghio S, Grunig E, Guazzi M, Kasprzak JD, Kolias T, Kovacs G, La Gerche A, Limogelli G, Marra AM, Matucci-Cerinic M, Mauro C, Moreo A, Pratali L, Ranieri B, Rega S, Rudski L, Saggar R, Salzano A, Serra W, Stanziola AA, Vannan MA, Voilliot D, Vriz O, Wierzbowska-Drabik K, Cittadini A, Naeije R, Bossone E; RIGHT Heart International NETwork (RIGHT-NET) Investigators. Exercise Stress Echocardiography of the Right Ventricle and Pulmonary Circulation. J Am Coll Cardiol. 2023 Nov 21;82(21):1973-1985. doi: 10.1016/j.jacc.2023.09.807. PMID 37968015